CLINICAL TRIAL: NCT02754297
Title: Personalized Peptide Receptor Radionuclide Therapy of Neuroendocrine Tumors: A Phase 2 Study
Brief Title: Personalized PRRT of Neuroendocrine Tumors
Acronym: P-PRRT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A14-11-2181
Record Dates: First submitted 2016-03-10; First posted 2016-04-28 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Neuroendocrine Tumors; Carcinoid Tumor; Carcinoma, Neuroendocrine
Keywords: Neuroendocrine tumors; Personalized; Peptide receptor radionuclide therapy; PRRT; 177Lu-DOTATATE; 177Lu-octreotate
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor; Carcinoma, Neuroendocrine | interventions — 177Lu-octreotate; lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Personalized PRRT (P-PRRT) (Experimental): 177Lu-Octreotate (LuTate) P-PRRT will be administered as follows:
  * Renal absorbed radiation dose will be prescribed for the 4-cycle induction course (23 Gy) and for each subsequent cycle (6 Gy), with a reduction in cases of impaired renal or bone marrow function, or significant toxicity from prior cycles.
  * The personalized activity to be administered at each cycle will be derived from renal dose per unit of injected activity that is predicted by patient characteristics or renal dose delivered during prior cycle(s).
  * Participants responding to the induction course of P-PRRT will be eligible to receive additional consolidation and/or maintenance cycles.
  * Participants with prior PRRT exposure outside the trial may receive less induction cycles, or only consolidation/maintenance cycle(s).
  Interventions: Drug: 177Lu-Octreotate

INTERVENTIONS:
Drug: 177Lu-Octreotate — * The induction course will consist in 4 cycles at 8-10 weeks intervals.
  * Concomitant amino acids will be administered for renal protection.
  * Intra-arterial LuTate administration will be allowed in suitable cases.
  * Dosimetry will be based on quantitative SPECT/CT imaging.
  * In patients with hormonal symptoms, somatostatine analogues can be given between P-PRRT cycles.
  Other Names: LuTate; 177Lu-[DOTA0,Tyr3]octreotate; 177Lu-DOTATATE

SUMMARY:
In this study, peptide receptor radionuclide therapy (PRRT) with 177Lu-Octreotate (LuTate) will be personalized, i.e. administered activity of LuTate will be tailored for each patient to maximize absorbed radiation dose to tumor, while limiting that to healthy organs.

The purpose of this study is to:

* Assess the objective (radiological), symptomatic and biochemical response rates following an induction course of personalized PRRT;
* Assess the overall, the disease-specific, and the progression-free survival following P-PRRT;
* Correlate therapeutic response and survival with tumor absorbed radiation dose;
* Evaluate the acute, subacute and chronic adverse events following P-PRRT;
* Correlate toxicity (i.e. occurence and severity of adverse events) with absorbed radiation doses to organs at risk;
* Optimize the quantitative SPECT imaging-based dosimetry methods in a subset of 20 patients (sub-study funded by the Canadian Institutes of Health Research).

This study also has a compassionate purpose, which is to provide access to PRRT to patients.

DETAILED DESCRIPTION:
A prospective, single-center, non-comparative, open phase 2 study. In this study, personalized peptide receptor radionuclide therapy (P-PRRT) with 177Lu-Octreotate (LuTate) will be administered to patients with progressive and/or symptomatic inoperable neuroendocrine tumors (NET) of any origin expressing the somatostatin receptor.

The primary objective to assess the objective response rate at 3 months following a four-cycle induction course of P-PRRT will be assessed for at least the first 85 participants.

This study as a compassionate aim to provide access to personalized PRRT patients at CHU de Québec - Université Laval center, and therefore this study has no pre-determined recruitment period duration or limited number of participants, and may remain open as long as necessary to fulfill this aim.

The study will continue until all participants have completed a minimum follow-up of 5 years. Interim analyses will be conducted annually.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from a progressive and/or symptomatic NET (any site);
* Patient ineligible to, or refusing a potentially curative treatment such as surgical resection;
* Patient who did not respond, is intolerant or refuses other indicated and available palliative treatments;
* Demonstration of overexpression of somatostatin receptor by tumor lesions by scintigraphic imaging (Octreoscan or 68Ga positron emission tomography.

Exclusion Criteria:

* Pregnancy;
* Breastfeeding;.
* Very limited survival prognosis (i.e. less than a few weeks, because of the NET disease or any other condition) or Eastern Cooperative Oncology Group (ECOG) 4 performance status;
* Inability to obtain informed consent of the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2025-04-12 (Estimated); Study Completion 2029-04-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3 months after induction course
  Primary efficacy endpoint is the objective response rate on contrast-enhanced CT (or MRI) by RECIST criteria (and secondarily by South Western Oncology Group (SWOG) criteria) at 3 months after the 4th induction cycle of P-PRRT, in comparison to pre-treatment scan (within 3 months before commencing P-PRRT).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Time from first cycle to date of disease progression or death, reported up to 5 years after accrual closure
  Progression of disease is defined as the time from first cycle to the date of first documented progression of disease or death due to any cause. Progression of disease is defined by RECIST criteria.
Overall survival (OS) | Time from first cycle to date of death, reported up to 5 years after accrual closure
Symptomatic response rate | 3 months after induction course
  Proportion of participants with improved, stable or worsened NET-related symptoms (frequency and severity), based on participant interviews at baseline and 3 months after completion of induction course.
Quality of life response | 3 months after induction course
  Proportion of participants with improved, stable or worsened quality of life score by EORTC quality of life questionnaires QLQ-C30 and QLQ-GI.NET21, administered at baseline and 3 months after induction course.
Biochemical response | 3 months after induction course
  Proportion of participants with improved (decreased by 25% or more), stable or worsened (increased by 25% or more) Chromogranin-A serum levels performed at baseline and 3 months after induction course.
Safety determined by type, frequency and severity of adverse events per CTCAE version 4.03 and type, frequency and severity of laboratory toxicities per CTCAE version 4.03 | From the first treatment cycle administration until 5 years after accrual closure or death, whichever came first

OTHER OUTCOMES:
Tumor radiation dose-response relationship | 3 months after induction course
  Correlation between cumulative absorbed radiation dose to tumor lesions and 3-month objective response rate, as defined above
Tumor radiation dose-survival relationship | At least 5 years after first cycle or until study completion, whichever came first
  Correlation between cumulative absorbed radiation dose to tumor lesions and survival endpoints above (PFS and OS)
Renal radiation dose-chronic toxicity relationship | At least 5 years after first cycle or until study completion, whichever came first
  Correlation between cumulative absorbed radiation dose to kidney and variations in glomerular filtration rate from baseline, reported annually for at least 5 years after first cycle or until study completion.
Bone marrow radiation dose-chronic toxicity relationship | At least 5 years after first cycle or until study completion, whichever came first
  Correlation between cumulative absorbed radiation dose to bone marrow and chronic variations of blood counts from baseline, reported annually for at least 5 years after first cycle or until study completion.
Bone marrow radiation dose-subacute toxicity relationship | Time of nadir blood counts values between 2 and 6 weeks after each cycle
  Correlation between per-cycle absorbed radiation dose to bone marrow and subacute variations (nadir values between 2 and 6 weeks) of blood counts from baseline, for each cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Mathieu Beauregard, MD,MSc,FRCPC, Principal Investigator — CHU de Québec - Université Laval
Locations (1):
- CHU de Québec - Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Del Prete M, Buteau FA, Arsenault F, Saighi N, Bouchard LO, Beaulieu A, Beauregard JM. Personalized 177Lu-octreotate peptide receptor radionuclide therapy of neuroendocrine tumours: initial results from the P-PRRT trial. Eur J Nucl Med Mol Imaging. 2019 Mar;46(3):728-742. doi: 10.1007/s00259-018-4209-7. Epub 2018 Nov 30. PMID 30506283